CLINICAL TRIAL: NCT02525224
Title: Nutritional Supplement Efficacy on Cellular Protection and Skin Health in Generally Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Collaborators: Dermatology Consulting Services, High Point NC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-PHX-0001; DCS-50-15 (Other: Dermatology Consulting Services)
Record Dates: First submitted 2015-08-13; First posted 2015-08-17 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Skin Health
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutritional Supplement (Other): Proprietary nutritional supplement
  Interventions: Dietary Supplement: Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement — 2 Hard-shell liquid capsules taken twice daily with breakfast and dinner.

SUMMARY:
Healthy skin has been equated with a healthy diet leading to the "inside out" approach to skin health. Since the skin is the barrier to the external world, healthy skin should lead to overall better health. Conversely, the skin derives its nutrition from the internal body requiring the consumption of nutritional supplements for optimal health. This research attempts to examine skin attributes and improved appearance achieved after consumption of a state-of-the-art dietary supplement.

DETAILED DESCRIPTION:
Subjects will present to the research center and complete an informed consent. They will undergo assessment for inclusion/exclusion criteria, skin examination, BMI calculation, and a brief medical history. Subjects that are found to be appropriate for study entry will undergo an investigator and subject facial evaluation. In addition, they will undergo noninvasive measurements of TEWL, corneometry, skin elasticity, dermspectrophotometry, and assessment with a biophotonic scanner. Facial photography will also be performed. A target site on the right or left sun protected buttock will be selected and will receive 1, 2, and 3 MED of solar simulated radiation.

Subjects will return to the research center 24 hours after irradiation for photography and erythema scaledermospectrophotometer measurement of the irradiated sites and biopsy of the 2 - 3 MED sites. The MED biopsy site will be consistent for each subject, but will be chosen based on the amount of achieved erythema. A 2mm punch biopsy will be taken of the irradiated site and another adjacent nonirradiated site for a total of 2 skin biopsies that will be closed with 5-0 nylon sutures. The biopsy from the nonirradiated site will be processed and shipped as instructed by the sponsor to a laboratory for epigenetic analysis. All subjects will be dispensed the supplement in a white bottle with a research center label along with a compliance diary. Subjects will return in 2 weeks just for suture removal.

At week 4, subjects will undergo an investigator and subject facial evaluation. In addition, they will undergo noninvasive measurements of TEWL, corneometry, skin elasticity, dermspectrophotometry, and assessment with a biophotonic scanner. Subjects will be redispensed study supplements.

Subjects will return to the research facility at week 8 and undergo noninvasive measurements of TEWL, corneometry, skin elasticity, dermspectrophotometry, and assessment with a biophotonic scanner. A target site on the right or left sun protected buttock will be selected and will receive 1, 2, and 3 MED of solar simulated radiation. All supplement bottles and unused product will be collected. Subjects will return to the research center 24 hours after irradiation for photography and erythema scale dermospectrophotometer measurement of the irradiated sites and biopsy of the 2-3 MED sites. The biopsy site will be the same MEDs as the original biopsy site at baseline. A 2mm punch biopsy will be taken of the irradiated site and another adjacent nonirradiated site for a total of 2 skin biopsies that will be closed with 5-0 nylon sutures. The biopsy from the nonirradiated site will be processed and shipped as instructed by the sponsor to a laboratory for epigenetic analysis. All supplement bottles and unused product will be collected. All bottles and unused product will be returned to the sponsor.

Subjects will return to the research center at week 10 for suture removal only.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be between 40-75 years of age with no known medical conditions that, in the investigator's opinion, may interfere with study participation.
* Individuals must present with moderate signs of aging
* Subject is willing and able to participate in all aspects of the study
* Individuals must sign informed consent, photo release consent and confidentiality agreement
* Subject eats 1 or less servings of fatty fish per week
* Subject has a BMI > 19 and < 30
* Subjects who have been on a stable dose of chronic use medications for at least 3 months prior to study participation
* Subjects who, in the opinion of the investigator, are free of any medical condition(s) that might affect study measures

Exclusion Criteria:

* Subject failure to provide informed consent
* Individuals that are being treated for cancer or have a history of facial skin cancer on the test areas
* Individuals with sunburn, moderate to pronounced suntan, even skin tones, tattoos, scars or other disfiguration, dilated vessels or other conditions on the test area that might influence the test results
* Any disease or condition of the skin that the examining investigator deems inappropriate for participation, including rosacea, eczema, psoriasis, and atopic dermatitis
* Individuals currently taking medications which in the opinion of the investigators may interfere with the study. This would include but not be limited to routine high dosage use of anti-inflammatory drugs (aspirin, ibuprofen, corticosteroids) immunosuppressive drugs or antihistamine medications (steroid nose drops and/or eye drops are permitted), and insulin, antibiotics or other topical drugs at the test sites.
* Individuals with uncontrolled metabolic diseases such as diabetes (Type I and II), hypertension, hyperthyroidism or hypothyroidism, severe chronic asthma, immunological disorders such as HIV positive, AIDS and systemic lupus erythematosus or mastectomy for cancer involving removal of lymph nodes
* Subject is taking supplemental oral dietary/nutritional supplements containing more than 800 IU of vitamin D, 200 mg fish oil, 200 mg krill oil, 2 mg total carotenoids (lycopene, lutein, etc.) and/or 5 mg resveratrol within 30 days prior to study product administration
* Difficulty in swallowing capsules
* Women known to be pregnant, nursing or planning to become pregnant
* Individuals participating in other facial clinical studies
* Individuals who have routinely used an alpha-hydroxyl-acid (AHA) or a beta-hydroxyl-acid (BHA) containing product within two weeks or Retin-A®, Retin-A Micro®, Renova®, Differin®, Avita®, Tazorac®, or Soriatane® within one month of the study start or have taken Accutane® within one year of the study start. Individuals who have used Retinol in the last six months
* Individuals with inflammatory acne lesions (i.e., papules, pustules, cysts, nodules) at the test site
* Individuals who have had chemical peels or dermabrasion within the last six months
* Individuals with known allergies to fish oil. Individuals currently using topically applied prescription medications where the medication is applied on or near the test site
* Individuals who have sun tanned (sun or tanning beds) in the nude within the past 1 year
* Excessive alcohol use (>2 drinks per day)
* Subject is a current smoker or quit less than 3 years from screening visit
* History of substance abuse
* Use of anti-aging treatment skin care products within 30 days of study enrollment and throughout study participation

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Cellular protection of the skin | 8 weeks
  The primary efficacy endpoint is to determine the effects of a nutritional supplement on cellular protection of the skin induced by UV radiation in generally healthy adults as determined by a reduction in sunburn cell count following supplement ingestion for 8 weeks.

SECONDARY OUTCOMES:
Skin Health | 8 weeks
  The secondary efficacy endpoint is to assess improvement in skin health characteristics in subjects consuming a dietary supplement as evidenced by improvement in the dermatologist investigator overall visual assessment of lines/wrinkles, firmness/elasticity, radiance, skin texture/smoothness, and overall appearance.

CONTACTS AND LOCATIONS:
Overall Officials: Zoe D Draelos, MD, Principal Investigator — Dermatology Consulting Services, High Point NC
Locations (1):
- Dermatology Consulting Services, High Point, North Carolina, United States